CLINICAL TRIAL: NCT02896179
Title: The Effects of an Innovative Combined Virtual Reality and Robot Assisted Gait Training on Cognitive and Walking Functions in Patients With Multiple Sclerosis: A Randomized Control Trial
Brief Title: Virtual Reality and Robot Assisted Gait Training in Patients With Multiple Sclerosis
Acronym: GE-O-VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Full Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE-O-VR
Record Dates: First submitted 2016-08-30; First posted 2016-09-12 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Gait rehabilitation; Quality of life; Virtual reality; Cognitive deficit; Robot assisted gait training
MeSH Terms: conditions — Multiple Sclerosis; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot-assisted gait training group+VR (Experimental): The first group will be subjected to Robot-assisted gait training (RAGT) for 6 weeks (2 sessions/ week) with a total of 12 sessions by mean of GEO System plus Virtual Reality scenario. During each session, the patients will practice 15 to 20 min of simulated floor walking with simulating of a real walking trail. Each session will last up to 50 minutes, the first 30 minutes will be dedicated to gait training and the last 20 minutes to stretch the lower limb's muscles.
  Interventions: Device: Robot-assisted gait training group+VR
- Robot-assisted gait training group (Active Comparator): The second group will be subjected to Robot-assisted gait training (RAGT) for 6 weeks (2 sessions/ week) with a total of 12 sessions by mean of GEO System. During each session, the patients will practice 15 to 20 min of simulated floor walking. Each session will last up to 50 minutes, the first 30 minutes will be dedicated to gait training and the last 20 minutes to stretch the lower limb's muscles.
  Interventions: Device: GEO

INTERVENTIONS:
Device: Robot-assisted gait training group+VR — The first group will be subjected to Robot-assisted gait training (RAGT) for 6 weeks (2 sessions/ week) with a total of 12 sessions by mean of GEO System plus Virtual Reality scenario. During each session, the patients will practice 15 to 20 min of simulated floor walking with simulating of a real walking trail. Each session will last up to 50 minutes, the first 30 minutes will be dedicated to gait training and the last 20 minutes to stretch the lower limb's muscles.
  Arms: Robot-assisted gait training group+VR
Device: GEO — The second group will be subjected to Robot-assisted gait training (RAGT) for 6 weeks (2 sessions/ week) with a total of 12 sessions by mean of GE-O System. During each session, the patients will practice 15 to 20 min of simulated floor walking. Each session will last up to 50 minutes, the first 30 minutes will be dedicated to gait training and the last 20 minutes to stretch the lower limb's muscles
  Arms: Robot-assisted gait training group

SUMMARY:
Multiple Sclerosis (MS), the most common non-traumatic cause of neurologic disability in young adults, affects mobility and ambulation in the majority of patients. Nearly 50% of persons with MS will require an assistive device to ambulate within 10 years of diagnosis. A subgroup of MS is Primary Progressive MS, which manifests with gait disturbances over 80% of patients in the long term. In addition to altered gait, nearly 70% of patients will experience cognitive deficits during the course of the disease. Therefore, actions that facilitate patient involvement in finding solutions for personalized management of disease and disability are needed.

Although immunomodulatory drugs offer some benefit in other types of Multiple Sclerosis, there is currently no effective treatment for Primary Progressive MS. A fundamental goal in the management of persons with MS is to maximize their ability to ambulate and perform safe and effective transfers in everyday life.

In the last decade, research has increasingly centered on the effects of robot devices in the rehabilitation of patients with neurological diseases. This has led to the development of new robot-assisted gait devices engendered by virtual-reality systems, and several studies have demonstrated the positive effects that these devices have on gait endurance and quality of life in patients with neurological diseases and disability.

The aim of this project is to develop and study the effects of a novel, cognitively intensive virtual-reality -based rehabilitation software application that simulates a real-world environment where a person can walk. The virtual-reality application is an upgrade version synchronized to a robotic device, the GEO System. The second aim is to compare the cognitive and motor effects of robot-assisted gait training with this application against training with robot-assisted gait training without virtual reality.

The experimental group will receive robot-assisted gait training with the virtual-reality application and the control group will receive robot-assisted gait training All subjects will undergo training for 6 weeks (2 sessions/week) for a total of 12 sessions. Assessments before training, after training, and at follow-up will be performed using clinical and instrumental tests to compare the effects of training.

Successful completion of the study may help patients to alleviate the impact of disability, increase their independence in activities of daily life, and improve their quality of life. Through new rehabilitative strategies that combine cognitive and motor training involving higher brain functions and motivation, patients will be stimulated to walk in a reality-based environment.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale between 3 and 6;
* Mini Mental Examination State >24;
* age >18 years;
* ability to sit without trunk support;
* ability to stand for at least 10 seconds with support;
* no botulinum toxin injection into the affected leg muscles or rehabilitation treatment in the 6 months before recruitment.

Exclusion Criteria:

* patients with disease recurrence that has worsened significantly during the 8 weeks before recruitment;
* changes in pharmacological therapy that could modify the disease course in the previous 3 months before recruitment;
* changes in pharmacological therapy for fatigue treatment in the previous 3 months before recruitment
* medications altering central nervous system (excitability (e.g., antiepileptics, neuroleptics, benzodiazepines or antidepressants) or with presumed effects on central nervous system plasticity (e.g., dopamine, fluoxetine or D-amphetamine);
* other neurological or orthopedic conditions involving the lower limbs (musculoskeletal diseases, severe osteoarthritis, peripheral neuropathy, joint replacement);
* cardiovascular co-morbidity (recent myocardial infarction, heart failure, uncontrolled hypertension, orthostatic hypotension).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
10 meters Walking test (10-MtWT) change in gait speed (m/sec) | Baseline time 0 and up to 12 weeks
  the test has been selected as a measure of gait speed. This is a validated test requiring individuals to walk on a flat hard floor at their fastest speed for 10 meters. Scoring is walking speed.

SECONDARY OUTCOMES:
Berg Balance Scale | Baseline time 0 and up to 12 weeks
2-Minute Walking Test (meters) | Baseline time 0 and up to 12 weeks
Activities-specific Balance Confidence Scale | Baseline time 0 and up to 12 weeks
Tower of London - point | Baseline time 0 and up to 12 weeks
  Tower of London assesses deficits in planning abilities and strategic problem solving. Two pictures are shown to the subject. Each picture shows three different colored balls arranged in different positions on three pegs. The subject has to transpose the three balls, starting from an initial position, to reach various final positions in a specific number of moves. The task comprises 12 problems with different target positions. For each problem, the participant earns three points if a solution is reached in only one attempt, two points if the solution is reached in two attempts, one point if the solution is reached in three attempts, and zero points if the solution is not reached in three attempts (range 0-36; higher scores=better performance)
Multiple Sclerosis Quality Of Life-54 | Baseline time 0 and up to 12 weeks
Gait Analysis - Cadence (step/min) | Baseline time 0 and up to 12 weeks
  It is an electronic system used for the gathering of the temporal-spatial data of deambulation. It is made up of an 8 meter long walkway connected to a computer. The system records the signal, reproducing the pressure maps of each step on video, identifying the progression of the center of gravity and recording all of the temporal-spatial features of gait.
Gait Analysis - Stride length (cm) | Baseline time 0 and up to 12 weeks
  It is an electronic system used for the gathering of the temporal-spatial data of deambulation. It is made up of an 8 meter long walkway connected to a computer. The system records the signal, reproducing the pressure maps of each step on video, identifying the progression of the center of gravity and recording all of the temporal-spatial features of gait.
Gait Analysis - Step length (cm) | Baseline time 0 and up to 12 weeks
  It is an electronic system used for the gathering of the temporal-spatial data of deambulation. It is made up of an 8 meter long walkway connected to a computer. The system records the signal, reproducing the pressure maps of each step on video, identifying the progression of the center of gravity and recording all of the temporal-spatial features of gait.
Gait Analysis - distance of heel to heel (cm) | Baseline time 0 and up to 12 weeks
  It is an electronic system used for the gathering of the temporal-spatial data of deambulation. It is made up of an 8 meter long walkway connected to a computer. The system records the signal, reproducing the pressure maps of each step on video, identifying the progression of the center of gravity and recording all of the temporal-spatial features of gait.
Gait Analysis - time of stance (sec) | Baseline time 0 and up to 12 weeks
  It is an electronic system used for the gathering of the temporal-spatial data of deambulation. It is made up of an 8 meter long walkway connected to a computer. The system records the signal, reproducing the pressure maps of each step on video, identifying the progression of the center of gravity and recording all of the temporal-spatial features of gait.
Gait Analysis - time of swing (sec) | Baseline time 0 and up to 12 weeks
  It is an electronic system used for the gathering of the temporal-spatial data of deambulation. It is made up of an 8 meter long walkway connected to a computer. The system records the signal, reproducing the pressure maps of each step on video, identifying the progression of the center of gravity and recording all of the temporal-spatial features of gait.
Gait Analysis - time of single support (sec) | Baseline time 0 and up to 12 weeks
  It is an electronic system used for the gathering of the temporal-spatial data of deambulation. It is made up of an 8 meter long walkway connected to a computer. The system records the signal, reproducing the pressure maps of each step on video, identifying the progression of the center of gravity and recording all of the temporal-spatial features of gait.
Gait Analysis - time of double support (sec) | Baseline time 0 and up to 12 weeks
  It is an electronic system used for the gathering of the temporal-spatial data of deambulation. It is made up of an 8 meter long walkway connected to a computer. The system records the signal, reproducing the pressure maps of each step on video, identifying the progression of the center of gravity and recording all of the temporal-spatial features of gait.
Body's Centre of Pressure length (mm) | Baseline time 0 and up to 12 weeks
  the static balance will be carried out with a monaxial platform, an electronic system used for the evaluation of the length of the centre of pressure (CoP)
Body's Centre of Pressure Area Path (mm2) | Baseline time 0 and up to 12 weeks
  the static balance will be carried out with a monaxial platform, an electronic system used for the evaluation of the length of the centre of pressure (CoP)
Sustained Attention to Response Task - Time of reaction time | Baseline time 0 and up to 12 weeks
  evaluates sustained attention, response inhibition, and reaction time. It is a go-no go target detection task composed of a series of numbers containing different digits from 1 to 9. The subject has to respond as quickly as possible to the appearance of each number by pressing a button, except when the number is 3. The score is the reaction times averaged over the test, and the total number of correct and incorrect responses
Phonemic Fluency Test | Baseline time 0 and up to 12 weeks
Paced Auditory Serial Addition Test | Baseline time 0 and up to 12 weeks
Trail Making Test | Baseline time 0 and up to 12 weeks
Wechsler Adult Intelligence Scale | Baseline time 0 and up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Smania, MD, Principal Investigator — Neuromotor and Cognitive Rehabilitation Center Department of Neurological and Movement Sciences University of Verona, Verona, Italy P.zza L.A. Scuro, 10 37134 Verona, Italia
Locations (1):
- Azienta Ospedaliera, SSO Rehabilitation Unit, Verona, Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No